CLINICAL TRIAL: NCT00300469
Title: A Multicenter, Randomized, Double-Blind, Prospective Study Comparing the Safety and Efficacy of Fenofibric Acid and Atorvastatin Calcium Combination Therapy to Fenofibric Acid and Atorvastatin Calcium Monotherapy in Subjects With Mixed Dyslipidemia
Brief Title: Evaluate Safety and Efficacy of ABT-335 in Combination With Atorvastatin in Subjects With Multiple Abnormal Lipid Levels in the Blood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-750
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Mixed Dyslipidemia; Coronary Heart Disease; Dyslipidemia
Keywords: Mixed Dyslipidemia; Coronary Heart Disease; Dyslipidemia
MeSH Terms: conditions — Coronary Disease; Dyslipidemias | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Active Comparator): ABT-335 + 20 mg atorvastatin
  Interventions: Drug: ABT-335; Drug: Atorvastatin
- B (Active Comparator): ABT-335 + 40 mg atorvastatin
  Interventions: Drug: ABT-335; Drug: Atorvastatin
- C (Placebo Comparator): ABT-335 monotherapy
  Interventions: Drug: ABT-335; Drug: Placebo
- D (Placebo Comparator): 20 mg atorvastatin monotherapy
  Interventions: Drug: Atorvastatin; Drug: Placebo
- E (Placebo Comparator): 40 mg atorvastatin monotherapy
  Interventions: Drug: Atorvastatin; Drug: Placebo
- F (Placebo Comparator): 80 mg atorvastatin monotherapy
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: ABT-335 — 135 mg, daily, 12 weeks
  Arms: A; B; C
Drug: Atorvastatin — Daily, 12 weeks, see Arm Description for dosage information
  Arms: A; B; D; E; F
Drug: Placebo — daily, 12 weeks, see Arm Description for placebo information
  Arms: C; D; E; F

SUMMARY:
The purpose of this study is to compare the safety and efficacy of fenofibric acid (ABT-335) + atorvastatin combination therapy with ABT-335 and atorvastatin monotherapy in subjects with multiple abnormal lipid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mixed dyslipidemia
* Subjects must agree to utilize adequate birth control methods and to adhere to the American Heart Association (AHA) diet

Exclusion Criteria:

* Subjects with unstable medical conditions or medical conditions considered inappropriate in a clinical trial.
* Patients who are taking certain medications or unstable dose of specific medications.
* Women who are pregnant or plan on becoming pregnant, or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2006-03; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Global Medical Information, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Bays HE, Roth EM, McKenney JM, Kelly MT, Thakker KM, Setze CM, Obermeyer K, Sleep DJ. The effects of fenofibric acid alone and with statins on the prevalence of metabolic syndrome and its diagnostic components in patients with mixed dyslipidemia. Diabetes Care. 2010 Sep;33(9):2113-6. doi: 10.2337/dc10-0357. Epub 2010 Jun 23. PMID 20573750
- [Derived] Jones PH, Cusi K, Davidson MH, Kelly MT, Setze CM, Thakker K, Sleep DJ, Stolzenbach JC. Efficacy and safety of fenofibric acid co-administered with low- or moderate-dose statin in patients with mixed dyslipidemia and type 2 diabetes mellitus: results of a pooled subgroup analysis from three randomized, controlled, double-blind trials. Am J Cardiovasc Drugs. 2010;10(2):73-84. doi: 10.2165/10061630-000000000-00000. PMID 20136164
- [Derived] Jones PH, Bays HE, Davidson MH, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Evaluation of a new formulation of fenofibric acid, ABT-335, co-administered with statins : study design and rationale of a phase III clinical programme. Clin Drug Investig. 2008;28(10):625-34. doi: 10.2165/00044011-200828100-00003. PMID 18783301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects were randomized but never treated: 2 were randomized but were deemed ineligible, 1 had a history of allergic reactions to statins, and 1 was noncompliant and never received study drug.
Groups:
- ABT-335 + 20 mg Atorvastatin: ABT-335 + 20 mg atorvastatin combination therapy once daily
- ABT-335 + 40 mg Atorvastatin: ABT-335 + 40 mg atorvastatin combination therapy once daily
- ABT-335: ABT-335 monotherapy once daily
- 20 mg Atorvastatin: 20 mg atorvastatin monotherapy once daily
- 40 mg Atorvastatin: 40 mg atorvastatin monotherapy once daily
- 80 mg Atorvastatin: 80 mg atorvastatin monotherapy once daily
Period: Overall Study
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Started | 110 (For all arms, "started" means treated.) | 110 | 112 | 113 | 109 | 55
Completed | 89 | 89 | 95 | 104 | 95 | 46
Not Completed | 21 | 21 | 17 | 9 | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin | Total
Number analyzed (Participants) | 110 | 110 | 112 | 113 | 109 | 55 | 609
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 87 | 83 | 95 | 93 | 87 | 44 | 489
  >=65 years | 23 | 26 | 17 | 20 | 22 | 11 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 57 | 48 | 60 | 29 | 311
  Male | 54 | 49 | 55 | 65 | 49 | 26 | 298
Region of Enrollment [Number; unit: participants]
  North America | 110 | 110 | 112 | 113 | 109 | 55 | 609

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Triglycerides From Baseline to Final Visit
Description: [(Week 12 triglycerides minus baseline triglycerides)/baseline triglycerides] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline triglyceride value and at least 1 postbaseline triglyceride value, last observation carried forward (excluding one subject with an extreme outlying value)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 105 | 102 | 104 | 108 | 105 | 52
percent change | -45.6 (3.36) | -42.1 (3.40) | -29.6 (3.35) | -16.5 (3.31) | -23.2 (3.35) | -30.4 (4.70)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Atorvastatin vs 20 mg Atorvastatin; An n = 92 per arm would provide >99% power to detect a 20% decrease in triglycerides relative to statin monotherapy for each combo therapy dose, assuming an SD of 30%; Test type: Superiority or Other; p < 0.001, ANCOVA — alpha = 0.05, all 3 primary endpoints had to show superiority of combo therapy in order to declare combo therapy successful at a given statin dose, Hochberg method for multiple comparison adjustment for 2 statin doses
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Atorvastatin vs 40 mg Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Final Visit
Description: [(Week 12 HDL-C minus baseline HDL-C)/baseline HDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline HDL-C value and at least 1 postbasline HDL-C value, last observation carried forward (excluding 1 subject with extreme outlying value)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 95 | 91 | 93 | 101 | 92 | 50
percent change | 14.0 (2.02) | 12.6 (2.08) | 19.9 (2.04) | 6.3 (1.96) | 5.3 (2.05) | 6.2 (2.75)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Atorvastatin vs 20 mg Atorvastatin; An n = 92 per arm would provide 99% power to detect a 13% increase in HDL-C relative to statin monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Atorvastatin vs 40 mg Atorvastatin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.010, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Final Visit
Description: [(Week 12 LDL-C minus baseline LDL-C)/baseline LDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline LDL-C value and at least 1 postbaseline LDL-C value, last observation carried forward (excluding 1 subject with extreme outlying value)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 97 | 96 | 97 | 103 | 95 | 50
percent change | -33.7 (1.91) | -35.4 (1.93) | -3.4 (1.90) | -37.1 (1.85) | -39.7 (1.92) | -46.0 (2.61)
Statistical Analysis 1: Comparison: ABT-335 + 20 mg Atorvastatin vs ABT-335; An n = 92 per arm would provide >99% power to detect a 31% decrease in LDL-C relative to ABT-335 monotherapy for each combo therapy dose, assuming an SD of 15%; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-335 + 40 mg Atorvastatin vs ABT-335; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Final Visit
Description: [(Week 12 non-HDL-C minus baseline non-HDL-C)/baseline non-HDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline non-HDL-C value and at least 1 postbaseline non-HDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 95 | 91 | 93 | 102 | 92 | 50
percent change | -40.8 (1.69) | -42.5 (1.74) | -14.8 (1.71) | -35.7 (1.64) | -41.7 (1.72) | -45.2 (2.30)

5. Secondary Outcome: Mean Percent Change in Very Low-density Lipoprotein Cholesterol (VLDL-C) From Baseline to Final Visit
Description: [(Week 12 VLDL-C minus baseline VLDL-C)/baseline VLDL-C] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline VLDL-C value and at least 1 postbaseline VLDL-C value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 103 | 101 | 104 | 107 | 105 | 52
percent change | -48.3 (3.72) | -53.5 (3.74) | -36.5 (3.66) | -26.2 (3.63) | -35.6 (3.66) | -38.9 (5.13)

6. Secondary Outcome: Mean Percent Change in Total Cholesterol From Baseline to Final Visit
Description: [(Week 12 total cholesterol minus baseline total cholesterol)/baseline total cholesterol] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline total cholesterol value and at least 1 postbaseline total cholesterol value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 105 | 102 | 104 | 109 | 105 | 52
percent change | -32.8 (1.32) | -34.6 (1.33) | -10.1 (1.32) | -29.6 (1.29) | -33.8 (1.31) | -38.2 (1.84)

7. Secondary Outcome: Mean Percent Change in Lipoprotein Apo B (Apo B) From Baseline to Final Visit
Description: [(Week 12 Apo B minus baseline Apo B)/baseline Apo B] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline ApoB value and at least 1 postbaseline ApoB value, LOCF
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 104 | 101 | 104 | 109 | 104 | 52
percent change | -37.0 (1.49) | -37.1 (1.52) | -12.4 (1.49) | -32.9 (1.46) | -35.3 (1.50) | -40.3 (2.08)

8. Secondary Outcome: Median Percent Change in High-sensitivity C-reactive Protein (hsCRP) From Baseline to Final Visit
Description: [(Week 12 hsCRP minus baseline hsCRP)/baseline hsCRP] x 100
Time Frame: Baseline to 12 Weeks (Final Visit)
Population: All randomized subjects with a baseline hsCRP value and at least 1 postbaseline hsCRP value, LOCF
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 104 | 101 | 104 | 109 | 104 | 52
percent change | -26.2 (24.76) [-49.7 to 0.3] | -42.9 (25.11) [-56.4 to -21.2] | -12.4 (24.65) [-41.2 to 42.8] | -29.6 (24.18) [-48.3 to 14.7] | -30.3 (25.08) [-51.7 to -2.4] | -31.9 (34.50) [-57.5 to -3.5]

ADVERSE EVENTS:
Arm/Group | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 1 | 2 | 3 | 2 | 2 | 2
Other Adverse Events (participants affected / at risk) | 50 | 50 | 50 | 45 | 57 | 33
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Coronary artery disease (Cardiac disorders) | 0/110 | 0/110 | 1/112 | 0/113 | 0/109 | 0/55
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0/110 | 0/110 | 0/112 | 1/113 | 0/109 | 0/55
Abdominal hernia (Gastrointestinal disorders) | 0/110 | 0/110 | 0/112 | 0/113 | 0/109 | 1/55
Crohn's disease (Gastrointestinal disorders) | 0/110 | 0/110 | 0/112 | 0/113 | 1/109 | 0/55
Cholecystitis (Hepatobiliary disorders) | 0/110 | 1/110 | 0/112 | 0/113 | 0/109 | 0/55
Cholelithiasis (Hepatobiliary disorders) | 0/110 | 1/110 | 0/112 | 0/113 | 0/109 | 0/55
Abscess jaw (Infections and infestations) | 0/110 | 0/110 | 0/112 | 0/113 | 1/109 | 0/55
Parotitis (Infections and infestations) | 0/110 | 0/110 | 0/112 | 0/113 | 1/109 | 0/55
Accidental overdose (Injury, poisoning and procedural complications) | 0/110 | 1/110 | 0/112 | 0/113 | 0/109 | 0/55
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0/110 | 0/110 | 0/112 | 0/113 | 0/109 | 1/55
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/110 | 0/110 | 1/112 | 0/113 | 0/109 | 0/55
Sciatica (Nervous system disorders) | 0/110 | 0/110 | 0/112 | 1/113 | 0/109 | 0/55
Syncope (Nervous system disorders) | 1/110 | 0/110 | 0/112 | 0/113 | 0/109 | 0/55
Deep vein thrombosis (Vascular disorders) | 0/110 | 0/110 | 1/112 | 0/113 | 0/109 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Atorvastatin | ABT-335 + 40 mg Atorvastatin | ABT-335 | 20 mg Atorvastatin | 40 mg Atorvastatin | 80 mg Atorvastatin
Abdominal pain upper (Gastrointestinal disorders) | 3/110 | 2/110 | 3/112 | 2/113 | 2/109 | 2/55
Constipation (Gastrointestinal disorders) | 3/110 | 4/110 | 1/112 | 2/113 | 1/109 | 1/55
Diarrhea (Gastrointestinal disorders) | 6/110 | 5/110 | 7/112 | 5/113 | 7/109 | 7/55
Dyspepsia (Gastrointestinal disorders) | 3/110 | 3/110 | 1/112 | 1/113 | 4/109 | 0/55
Nausea (Gastrointestinal disorders) | 5/110 | 8/110 | 4/112 | 2/113 | 6/109 | 4/55
Fatigue (General disorders) | 1/110 | 2/110 | 0/112 | 3/113 | 6/109 | 0/55
Edema peripheral (General disorders) | 2/110 | 0/110 | 2/112 | 0/113 | 7/109 | 2/55
Bronchitis (Infections and infestations) | 0/110 | 1/110 | 0/112 | 0/113 | 1/109 | 2/55
Gastroenteritis viral (Infections and infestations) | 0/110 | 1/110 | 1/112 | 0/113 | 1/109 | 3/55
Influenza (Infections and infestations) | 1/110 | 3/110 | 0/112 | 4/113 | 1/109 | 1/55
Nasopharyngitis (Infections and infestations) | 4/110 | 3/110 | 4/112 | 4/113 | 4/109 | 3/55
Sinusitis (Infections and infestations) | 2/110 | 5/110 | 3/112 | 2/113 | 2/109 | 1/55
Upper respiratory tract infection (Infections and infestations) | 4/110 | 3/110 | 9/112 | 2/113 | 6/109 | 0/55
Alanine aminotransferase increased (Investigations) | 6/110 | 1/110 | 1/112 | 0/113 | 0/109 | 2/55
Aspartate aminotransferase increased (Investigations) | 6/110 | 1/110 | 1/112 | 0/113 | 0/109 | 2/55
Blood alkaline phosphatase increased (Investigations) | 1/110 | 0/110 | 0/112 | 0/113 | 2/109 | 2/55
Blood creatine phosphokinase increased (Investigations) | 4/110 | 0/110 | 0/112 | 0/113 | 1/109 | 2/55
Hepatic enzyme increased (Investigations) | 4/110 | 5/110 | 1/112 | 0/113 | 1/109 | 1/55
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/110 | 2/110 | 6/112 | 2/113 | 6/109 | 1/55
Back pain (Musculoskeletal and connective tissue disorders) | 5/110 | 1/110 | 5/112 | 5/113 | 6/109 | 0/55
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4/110 | 4/110 | 3/112 | 4/113 | 4/109 | 1/55
Myalgia (Musculoskeletal and connective tissue disorders) | 2/110 | 5/110 | 3/112 | 5/113 | 8/109 | 3/55
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/110 | 3/110 | 2/112 | 4/113 | 6/109 | 2/55
Dizziness (Nervous system disorders) | 3/110 | 7/110 | 3/112 | 1/113 | 4/109 | 0/55
Headache (Nervous system disorders) | 13/110 | 10/110 | 14/112 | 17/113 | 14/109 | 7/55
Somnolence (Nervous system disorders) | 1/110 | 0/110 | 1/112 | 0/113 | 1/109 | 2/55
Insomnia (Psychiatric disorders) | 1/110 | 1/110 | 3/112 | 1/113 | 2/109 | 2/55
Cough (Respiratory, thoracic and mediastinal disorders) | 1/110 | 1/110 | 2/112 | 2/113 | 1/109 | 3/55
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/110 | 5/110 | 3/112 | 4/113 | 4/109 | 0/55
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1/110 | 0/110 | 3/112 | 1/113 | 1/109 | 2/55
Pain (General disorders) | 4/110 | 4/110 | 3/112 | 1/113 | 1/109 | 2/55
Toothache (Gastrointestinal disorders) | 3/110 | 1/110 | 4/112 | 2/113 | 2/109 | 1/55
Vomiting (Gastrointestinal disorders) | 2/110 | 2/110 | 2/112 | 0/113 | 0/109 | 4/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall be so restricted after the expiration of twelve (12) months from completion of the studies at all sites. Any presentation or publication to be submitted to Sponsor (in draft of the same) for Sponsor review and comment.